CLINICAL TRIAL: NCT02601625
Title: A Randomized, Phase 1, Placebo-controlled, Double-blind, Single-dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Subcutaneously and Intravenously Delivered Anifrolumab in Healthy Subjects.
Brief Title: A Study to Assess the Pharmacokinetics and Safety of Single Doses of Anifrolumab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3461C00006
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Safety; Pharmacokinetics; Healthy Subjects
Keywords: Tolerability; Anifrolumab; Subcutaneous injection; Intravenous infusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Anifrolumab 300 mg SC injections (Experimental): 300 mg single dose anifrolumab delivered as 2 separate 1 mL SC injections administered serially
  Interventions: Drug: Anifrolumab SC injection (300mg)
- Anifrolumab 300 mg IV infusion (Experimental): 300 mg single dose anifrolumab delivered as an IV infusion over 30 minutes
  Interventions: Drug: Anifrolumab IV infusion (300mg)
- Anifrolumab 600 mg SC infusion (Experimental): 600 mg single dose anifrolumab or placebo delivered as 4 mL SC by infusion pump
  Interventions: Drug: Anifrolumab SC infusion (600mg)
- Placebo 300 mg SC injections (Placebo Comparator): 300 mg single dose placebo delivered as 2 separate 1 mL SC injections administered serially
  Interventions: Drug: Anifrolumab placebo SC injection (300mg)
- Placebo 300 mg IV infusion (Placebo Comparator): 300 mg single dose placebo delivered as an IV infusion over 30 minutes
  Interventions: Drug: Anifrolumab placebo IV infusion (300mg)
- Placebo 600mg SC infusion (Placebo Comparator): 600 mg single dose placebo delivered as 4 mL SC by infusion pump
  Interventions: Drug: Anifrolumab placebo SC infusion (600mg)

INTERVENTIONS:
Drug: Anifrolumab SC injection (300mg) — 300 mg of anifrolumab delivered as 2 separate 1 mL SC injections administered serially on Day 1
  Arms: Anifrolumab 300 mg SC injections
Drug: Anifrolumab IV infusion (300mg) — 300 mg of anifrolumab delivered as an IV infusion over 30 minutes on Day 1
  Arms: Anifrolumab 300 mg IV infusion
Drug: Anifrolumab SC infusion (600mg) — 600 mg of anifrolumab delivered as 4 mL SC by infusion pump on Day 1
  Arms: Anifrolumab 600 mg SC infusion
Drug: Anifrolumab placebo SC injection (300mg) — 300mg of placebo delivered as 2 separate 1 mL SC injections administered serially on Day 1
  Arms: Placebo 300 mg SC injections
Drug: Anifrolumab placebo IV infusion (300mg) — 600mg of placebo delivered as an IV infusion over 30 minutes on Day 1
  Arms: Placebo 300 mg IV infusion
Drug: Anifrolumab placebo SC infusion (600mg) — 600 mg of placebo delivered as 4 mL SC by infusion pump on Day 1
  Arms: Placebo 600mg SC infusion

SUMMARY:
This is a Phase I, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Pharmacokinetics and Safety of anifrolumab following Single-Dose administration to healthy subjects

DETAILED DESCRIPTION:
This is a Phase I placebo-controlled study to assess the pharmacokinetics, safety and tolerability of 2 doses of anifrolumab via the subcutaneous (SC) route of administration and 1 dose of anifrolumab via intravenous (IV) route in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 - 55 years.
3. Females must have a negative pregnancy test at screening.
4. Females with an intact cervix must have documentation of a Pap smear with no documented malignancy.
5. Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive, and weigh at least 50 kg.
6. Must have adequate abdominal adipose tissue for SC injection.
7. No history of latent or active TB prior to screening.
8. A chest radiograph with no evidence of current active infection or old active TB, malignancy, or clinically significant abnormalities within 6 months prior to screening.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which may put the subject at risk .
2. History or presence of hepatic or renal disease.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 8 weeks of participation .
4. Any clinically significant chronic or recent infection requiring hospitalization or treatment with anti-infectives.
5. History of cancer, apart from squamous or basal cell carcinoma of the skin.
6. Any clinically significant lab, vital sign or ECG abnormalities as judged by the investigator.
7. Known history of a primary immunodeficiency,HIV splenectomy or an underlying condition.
8. Any positive result on screening for hepatitis B, hepatitis C or HIV antibody.
9. History of drug abuse within 1 year of participation.
10. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 4 weeks or 5 half-lives prior to participation.
11. Previous receipt of:

    * Anifrolumab;
    * B cell-depleting therapy (including but not limited to epratuzumab, ocrelizumab, or rituximab) ≤ 52 weeks prior to screening.
12. History of allergy/hypersensitivity to drugs with a similar chemical structure or class to anifrolumab or to any human gamma globulin therapy.
13. Any live or attenuated vaccine within 8 weeks prior to participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit, Baltimore, United States of America
Locations (1):
- Research Site, Baltimore, Maryland, United States

REFERENCES:
- See also: d3461c00006-revised-study-protocol-1_REDACTED — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3872&filename=d3461c00006-revised-study-protocol-1_REDACTED.PDF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the PAREXEL Early Phase Clinical Unit Baltimore, 3001 S. Hanover St.
  Baltimore, MD 21225 United States of America
Pre-assignment Details: All eligible participants underwent a screening period of a maximum of 28 days. During the treatment period all participants were asked to be the residents at the study site prior to the evening meal the night before dosing with anifrolumab or placebo (Day -1) until at least 48 hours after dosing; and were then discharged on the morning of Day 3.
Groups:
- Anifrolumab 300 mg SC Injections: Participants received a single dose of anifrolumab 300 mg delivered as 2 separate 1 mL subcutaneous (SC) injections administered serially on Day 1.
- Anifrolumab 300 mg IV Infusion: Participants received single dose of anifrolumab 300 mg delivered as an intravenous (IV) infusion over 30 minutes on Day 1
- Anifrolumab 600 mg SC Infusion: Participants received single dose of anifrolumab 600 mg delivered as 4 mL SC by infusion pump on Day 1
- Pooled Placebo: Randomized participants received Anifrolumab matching placebo.
Period: Overall Study
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion | Pooled Placebo
Started (Participants) | 6 | 6 | 6 | 12
Completed (Participants) | 6 | 6 | 5 | 11
Not Completed | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Thirty healthy male and female subjects were included in this study, 6 subjects per anifrolumab treatment (300 mg anifrolumab SC, 300 mg anifrolumab IV, 600 mg anifrolumab SC) and 12 subjects for placebo treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion | Pooled Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (6.89) | 29.7 (7.97) | 26.3 (6.65) | 38.4 (12.26) | 32.1 (10.62)
Sex/Gender, Customized [Number; unit: Count of participants]
  Female | 4 | 1 | 2 | 4 | 11
  Male | 2 | 5 | 4 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Observed Maximum Serum Concentration (Cmax) Following Single Dose of Anifrolumab.
Description: To evaluate Cmax of anifrolumab after single administration of two doses subcutaneously and one dose intravenously.
  Up to 13 blood samples were collected in total.
Time Frame: On Day 1 pre-dose and at 5 minutes (IV cohort only), 24 and 48 hours post-dose and at each follow-up visit, up to 85 days
Population: The pharmacokinetic (PK) analysis set consisted of all participants in the safety analysis set for whom at least 1 of the primary PK parameters could be calculated, and who had no major protocol deviations that had an impact on the analysis of the PK data
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion
Number analyzed (Participants) | 6 | 6 | 6
ug/mL | 36.22 (11.63) | 82.44 (13.16) | 63.86 (20.45)

2. Primary Outcome: Pharmacokinetics: Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) Following Single Dose of Anifrolumab
Description: To evaluate AUC(0-t) of anifrolumab after single administration of two doses subcutaneously and one dose intravenously
  Up to 13 blood samples were collected in total.
Time Frame: as for outcome 1
Population: The PK analysis set consisted of all participants in the safety analysis set for whom at least 1 of the primary PK parameters could be calculated, and who had no major protocol deviations that had an impact on the analysis of the PK data
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion
Number analyzed (Participants) | 6 | 6 | 6
day*μg/mL | 769.1 (336.9) | 902.9 (175.8) | 1639 (557.7)

3. Primary Outcome: Pharmacokinetics: Area Under Serum Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC) Following Single Dose of Anifrolumab
Description: To evaluate AUC of anifrolumab after single administration of two doses subcutaneously and one dose intravenously.
  Up to 13 blood samples were collected in total.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion
Number analyzed (Participants) | 6 | 6 | 6
day*μg/mL | 784.6 (330.6) | 906.5 (174.9) | 1828 (679.8)

4. Primary Outcome: Safety: Number of Participants With Adverse Events (AEs)
Description: To assess the safety and tolerability of single doses of anifrolumab
Time Frame: From screening to final follow-up visit, up to 16 weeks
Population: The safety analysis set included all participants who received at least 1 dose of investigational medicinal product (IMP) (anifrolumab or placebo) and for whom any safety post-dose data were available.
Measure: Number; unit: Participants
Groups:
- Placebo 300 mg Anifrolumab SC: Participants received a single dose of placebo 300 mg delivered as 2 separate 1 mL subcutaneous (SC) injections administered serially on Day 1.
- Placebo 600 mg Anifrolumab SC: Participants received single dose of placebo 600 mg delivered as 4 mL SC by infusion pump.
- Placebo 300 mg Anifrolumab IV: Participants received Single dose of placebo 300 mg delivered as an IV infusion over 30 minutes.
- All Anifrolumab Participants: Overall number of participants who received anifrolumab therapy.
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion | Pooled Placebo | Placebo 300 mg Anifrolumab SC | Placebo 600 mg Anifrolumab SC | Placebo 300 mg Anifrolumab IV | All Anifrolumab Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4 | 4 | 4 | 18
Participants | 3 | 2 | 4 | 4 | 1 | 2 | 1 | 9

5. Primary Outcome: Safety: Summary of Local Injection Site Pain (SC Cohorts) Assessed in Participants
Description: Local injection site pain was assessed using a 100 mm participant rated Visual Analog Scale (VAS 0mm - 100mm ungraduated scale, where 0 = "no pain" to 100 = "worst imaginable pain"). This assessment was taken for only those participants in subcutaneously dosed treatment groups; 600 mg SC and 300 mg SC, anifrolumab and placebo. For the 300 mg SC anifrolumab and 300 mg SC placebo groups which received two simultaneous injections, the average VAS score (0mm-100mm) of the two injection sites were reported.
Time Frame: Immediately after dosing, at 10, 20 minutes and 1 hour after injection
Population: The safety analysis set included all participants who received at least 1 dose of IMP (anifrolumab or placebo) and for whom any safety post-dose data were available.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 600 mg SC Infusion | Placebo 300 mg Anifrolumab SC | Placebo 600 mg Anifrolumab SC
Number analyzed (Participants) | 6 | 6 | 4 | 4
Millimeter
  Immediately after dosing | 1.2 (2.21) | 0.0 (0.00) | 8.0 (13.69) | 0.0 (0.00)
  10 min after injection | 0.5 (0.63) | 0.0 (0.00) | 0.5 (1.00) | 0.0 (0.00)
  20 min after injection | 0.3 (0.42) | 0.0 (0.00) | 0.4 (0.75) | 0.3 (0.50)
  1 hour after injection | 0.2 (0.41) | 0.0 (0.00) | 0.3 (0.50) | 0.0 (0.00)

6. Primary Outcome: Safety: Summary of Local Injection Site Pruritus (SC Cohorts) Assessed in Participants
Description: Local injection site pruritus was assessed using a 100 mm participant rated Visual Analog Scale (VAS 0mm - 100mm ungraduated scale, where 0 = "no itching" to 100 = "worst imaginable itching"). This assessment was taken for only those participants in subcutaneously dosed treatment groups; 600 mg SC and 300 mg SC, anifrolumab and placebo. For the 300 mg SC anifrolumab and 300 mg SC placebo groups which received two simultaneous injections, the average VAS score (0mm-100mm) of the two injection sites were reported.
Time Frame: Immediately after dosing, at 10, 20 minutes and 1 hour after injection
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 600 mg SC Infusion | Placebo 300 mg Anifrolumab SC | Placebo 600 mg Anifrolumab SC
Number analyzed (Participants) | 6 | 6 | 4 | 4
Millimeter
  Immediately after dosing | 1.3 (2.60) | 14.0 (20.29) | 1.3 (1.66) | 0.8 (0.96)
  10 min after injection | 0.7 (1.21) | 6.3 (14.56) | 0.6 (1.25) | 0.0 (0.00)
  20 min after injection | 0.3 (0.52) | 1.5 (3.67) | 0.5 (1.00) | 0.3 (0.50)
  1 hour after injection | 0.1 (0.20) | 0.0 (0.00) | 0.4 (0.75) | 0.0 (0.00)

7. Primary Outcome: Safety: Summary of Erythema Injection Site Reaction (SC Cohorts) Assessed in Participants
Description: Erythema was measured as the largest diameter across the needle site on the skin in millimetres (mm). This assessment was taken for only those participants in subcutaneously dosed treatment groups; 600 mg SC and 300 mg SC, anifrolumab and placebo. For the 300 mg SC anifrolumab and 300 mg SC placebo groups which received two simultaneous injections, the average of the two injection site diameters (mm) were reported.
Time Frame: Immediately after dosing, at 10, 20 minutes and 1 hour after injection
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimeter
Groups:
- Placebo 300mg SC Injection: Participants received 300 mg single dose placebo delivered as 2 separate 1 mL SC injections administered serially on Day 1.
- Placebo 600 mg SC Injection: Participants received placebo 600mg
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 600 mg SC Infusion | Placebo 300mg SC Injection | Placebo 600 mg SC Injection
Number analyzed (Participants) | 6 | 6 | 4 | 4
Millimeter
  Immediately after dosing | 0.3 (0.42) | 17.0 (19.75) | 11.5 (14.62) | 20.0 (13.54)
  10 minutes after injection | 2.0 (4.18) | 17.5 (21.39) | 5.1 (9.59) | 18.0 (14.99)
  20 minute after injection | 2.7 (4.14) | 16.6 (20.81) | 5.5 (9.11) | 26.0 (18.55)
  1 hour after injection | 0.3 (0.52) | 2.5 (6.12) | 0.3 (0.50) | 10.0 (14.14)

8. Secondary Outcome: Evaluation of Immunogenicity of Anifrolumab IV Infusions and SC Injections by the Measurement of Anti-drug Antibody (ADA).
Description: Immunogenicity was assessed in all groups by the presence or absence of ADA, which was determined in serum samples using validated bioanalytical methods. The reported results are based on the confirmatory assay (positive/negative) of the ADA. The number of participants with positive, negative and missing results are reported for each time point using the safety analysis set.
Time Frame: Pre-dose and at Days 5 and Day 29, up to 85 days
Population: The safety analysis set included all subjects who received at least 1 dose of IMP (anifrolumab or placebo) and for whom any safety post-dose data were available.
Measure: Number; unit: Participants
Groups:
- All Subjects: Overall participants.
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Anifrolumab 600 mg SC Infusion | Pooled Placebo | All Subjects
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 30
Participants
  Day 1, pre-dose (positive) | 0 | 0 | 0 | 0 | 0
  Day 1, pre-dose (negative) | 6 | 6 | 6 | 12 | 30
  Day 1, pre-dose (missing) | 0 | 0 | 0 | 0 | 0
  Day 5 (positive) | 0 | 0 | 0 | 0 | 0
  Day 5 (negative) | 6 | 6 | 6 | 12 | 30
  Day 5 (missing) | 0 | 0 | 0 | 0 | 0
  Day 29 (positive) | 0 | 0 | 0 | 0 | 0
  Day 29 (negative) | 6 | 6 | 5 | 11 | 28
  Day 29 (missing) | 0 | 0 | 1 | 1 | 2
  Day 85 (positive) | 0 | 1 | 0 | 0 | 1
  Day 85 (negative) | 6 | 5 | 5 | 11 | 27
  Day 85 (missing) | 0 | 0 | 1 | 1 | 2

9. Primary Outcome: Safety: Summary of the Induration Injection Site Reaction (SC Cohorts) Assessed in Participants
Description: Induration was measured as the largest diameter across the needle site on the skin in millimetres (mm). This assessment was taken for only those participants in subcutaneously dosed treatment groups; 600 mg SC and 300 mg SC, anifrolumab and placebo. For the 300 mg SC anifrolumab and 300 mg SC placebo groups which received two simultaneous injections, the average of the two injection site diameters (mm) were reported.
Time Frame: Immediately after dosing, at 10, 20 minutes and 1 hour after injection
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 600 mg SC Infusion | Placebo 300mg SC Injection | Placebo 600 mg Anifrolumab SC
Number analyzed (Participants) | 6 | 6 | 4 | 4
Millimeter
  Immediately after dosing | 4.2 (10.21) | 22.5 (13.69) | 0.0 (0.00) | 12.5 (15.00)
  10 minutes after injection | 0.8 (2.04) | 17.3 (12.39) | 0.0 (0.00) | 16.5 (19.21)
  20 minute after injection | 0.1 (0.20) | 14.1 (11.41) | 0.1 (0.25) | 8.0 (16.00)
  1 hour after injection | 0.0 (0.00) | 11.7 (13.29) | 0.0 (0.00) | 12.5 (25.00)

ADVERSE EVENTS:
Time Frame: From screening to final follow-up visit, up to 16 weeks
Description: An adverse event (AE) is any undesirable medical condition or the deterioration of a pre existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Groups:
- Placebo 300 mg IV Infusion: Participants received 300 mg single dose placebo delivered as an IV infusion over 30 minutes on Day 1.
- Placebo 600 mg Anifrolumab (SC): Participants received 600 mg single dose placebo delivered as 4 mL SC by infusion pump on Day 1.
- All Anifrolumab Subjects: Overall number of participants who received anifrolumab therapy
Arm/Group | Anifrolumab 300 mg SC Injections | Anifrolumab 300 mg IV Infusion | Placebo 300 mg Anifrolumab SC | Placebo 300 mg IV Infusion | Placebo 600 mg Anifrolumab (SC) | Anifrolumab 600 mg SC Infusion | Pooled Placebo | All Anifrolumab Subjects
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/4 | 0/6 | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/4 | 0/6 | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 1/4 | 1/4 | 2/4 | 4/6 | 4/12 | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Anifrolumab 300 mg SC Injections (N=6) | Anifrolumab 300 mg IV Infusion (N=6) | Placebo 300 mg Anifrolumab SC (N=4) | Placebo 300 mg IV Infusion (N=4) | Placebo 600 mg Anifrolumab (SC) (N=4) | Anifrolumab 600 mg SC Infusion (N=6) | Pooled Placebo (N=12) | All Anifrolumab Subjects (N=18)
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1/4 | 0/1 | 0/1 | 0/2 | 0/1 | 0/2 | 0/4 | 1/7
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All of the study information and data collected during the study are confidential and the property of AstraZeneca. After completion of the study, the investigator may prepare a joint publication with AstraZeneca. The investigator must undertake not to submit any part of the individual data from this study for publication without prior consent of AstraZeneca at a mutually agreed time.